CLINICAL TRIAL: NCT07231354
Title: The Role of Physiotherapy in the Mental Health of Children and Adolescents With Neurodevelopmental Disorders: A Randomized Controlled Trial
Brief Title: Physiotherapy for Improving Mental Health in Children and Adolescents With ASD and ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Marianna Stavropoulou, Principal Investigator, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IHU-MST-2023-01
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder (ASD); Attention Deficit Hyperactivity Disorder (ADHD); Neurodevelopmental Disorders
Keywords: Physiotherapy; Mental Health; Children; Adolescents; Exercise Therapy; Rehabilitation
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Two-arm parallel-group randomized controlled design.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded to group assignment to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy Intervention Group (Experimental): Participants receive a structured physiotherapy program designed to improve emotional regulation, reduce anxiety symptoms, and enhance overall mental health. The program includes sensorimotor exercises, coordination training, postural activities, and structured physical activity tailored to children and adolescents with ASD or ADHD.
  Interventions: Behavioral: Structured Physiotherapy Program
- Comparator Group (No Intervention): Participants do not receive physiotherapy during the study period but continue their usual daily routines. After study completion, they are offered the physiotherapy program.

INTERVENTIONS:
Behavioral: Structured Physiotherapy Program — A structured multimodal physiotherapy program including sensorimotor integration exercises, balance and coordination training, postural control activities, therapeutic physical activity, breathing regulation techniques, and proprioceptive stimulation. The intervention is tailored to children and adolescents with ASD or ADHD and aims to improve emotional regulation, reduce anxiety, enhance behavioral self-control, and promote overall mental health.
  Arms: Physiotherapy Intervention Group

SUMMARY:
This study investigates whether a structured physiotherapy program can help reduce symptoms of stress, anxiety, and depression in children and adolescents diagnosed with Autism Spectrum Disorder (ASD) or Attention-Deficit/Hyperactivity Disorder (ADHD). ASD and ADHD are neurodevelopmental conditions often associated with emotional and behavioral challenges, including elevated levels of psychological distress.

The physiotherapy intervention includes techniques such as diaphragmatic breathing, acupressure, relaxation exercises, proprioceptive activities, and therapeutic positions designed to support emotional regulation. Children aged 6-18 years are randomly assigned to either an intervention group receiving the physiotherapy program or a control group receiving usual care.

The purpose of the study is to evaluate whether this physiotherapy protocol can positively influence emotional well-being and behavioral indicators related to ASD and ADHD. Outcomes are assessed using validated questionnaires measuring stress, anxiety, depression, and disorder-related behavioral characteristics before and after the intervention.

DETAILED DESCRIPTION:
This study examines the implementation of a structured physiotherapy program designed for children and adolescents diagnosed with Autism Spectrum Disorder (ASD) or Attention-Deficit/Hyperactivity Disorder (ADHD). The intervention includes breathing exercises, relaxation techniques, proprioceptive activities, and therapeutic postures aimed at supporting emotional regulation and reducing psychological distress.

Participants aged 6 to 18 years are randomly assigned to either an intervention group receiving the physiotherapy program or a control group receiving usual care. Standardized assessment tools are used to measure stress, anxiety, depression, and behavioral characteristics related to ASD and ADHD. The study follows a parallel-group randomized design and aims to evaluate the feasibility and potential therapeutic impact of physiotherapy-based approaches in this population.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) or Attention Deficit Hyperactivity Disorder (ADHD) by a qualified clinician.
* Age between 6 and 18 years.
* Ability to participate in structured physiotherapy sessions.
* Stable medication regimen (if applicable) for at least 4 weeks prior to study entry.
* Parent/guardian consent and child assent (where applicable).
* Ability of parents/guardians to comply with study procedures and assessments.

Exclusion Criteria:

* Severe intellectual disability that prevents participation in physiotherapy activities.
* Uncontrolled epilepsy or other neurological disorders that pose safety risks.
* Severe sensory or motor impairments preventing safe exercise participation.
* Participation in another clinical study within the last 3 months.
* Any acute medical condition deemed unsafe for physical activity.
* Behavioral issues that prevent structured participation (e.g., aggressive behavior).

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Stress Levels (DASS-21 Stress Subscale) | Baseline and post-intervention (after 10 sessions - approximately 5 weeks)
  Stress levels assessed using the DASS-21 Stress Subscale (score range 0-42). Higher scores indicate higher stress. The outcome will be analyzed as the change in score from baseline to post-intervention.
Change in Anxiety Levels (DASS-21 Anxiety Subscale) | Baseline and post-intervention (after 10 sessions - approximately 5 weeks)
  Stress/anxiety levels assessed using the DASS-21 Anxiety Subscale (score range 0-42). Higher scores indicate greater anxiety symptoms. The outcome will be analyzed as the change in score from baseline to post-intervention.
Change in Depression Levels (DASS-21 Depression Subscale) | Baseline and post-intervention (after 10 sessions - approximately 5 weeks)
  Depression levels assessed using the DASS-21 Depression Subscale (score range 0-42). Higher scores indicate higher depressive symptoms. The outcome will be analyzed as the change in score from baseline to post-intervention.

SECONDARY OUTCOMES:
Change in Autism-Related Behavioral Indicators (CAST Score) | Baseline and post-intervention (after 10 sessions - approximately 5 weeks)
  Assessment of autism-related behavioral characteristics using the CAST questionnaire (score range depends on the Greek validated version). Higher scores indicate greater autism-related behavioral traits. Outcome analyzed as the change in CAST score from baseline to post-intervention.
Change in ADHD-Related Behavioral Indicators (ADHD Parent Questionnaire Score) | Baseline and post-intervention (after 10 sessions - approximately 5 weeks)
  Assessment of ADHD-related behaviors using the ADHD Parent Questionnaire. Higher scores indicate more severe ADHD-related symptoms. Outcome analyzed as the change in score from baseline to post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Illias Kallistratos, Principal Investigator — International Hellenic University
Locations (1):
- Hippokratio General Hospital of Thessaloniki - Child Psychiatry Department, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Participant-level data will not be shared in order to protect confidentiality, as the dataset includes sensitive information from children and adolescents